CLINICAL TRIAL: NCT03445286
Title: Effect of Silver Diamine Fluoride on the Treatment of Gingivitis in Geriatric Patients
Brief Title: Silver Diamine Fluoride and Gingivitis in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A & M University Baylor College Of Dentistry (Other)
Responsible Party: Principal Investigator, Amal Noureldin, Clinical Associate Professor, Texas A & M University Baylor College Of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2017-0917
Record Dates: First submitted 2018-02-13; First posted 2018-02-26 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Gingivitis
Keywords: Gingivitis and geriatric patients; Silver Diamine Fluoride and gingivitis; Sliver Diamine Fluoride
MeSH Terms: conditions — Gingivitis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The participants with gingivitis are randomly allocated to two groups: group 1(case group) who will receive SDF application once every week within three weeks period and group 2 (control group) who will receive normal saline application once a week within three-week period
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and outcome Assessor will be blinded The participants will be blinded about which interventions they will receive and the Outcomes Assessor who will evaluate the gingival condition will be blinded about the interventions, and also the care provider who will apply the intervention will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Silver Diamine Fluordie Application (Experimental): This group will receive Silver Diamine Fluoride (SDF) application once every week within three weeks period
  Interventions: Device: Silver Diamine Fluoride
- Normal Saline (Placebo Comparator): This control group will receive normal saline application once a week within a a three-week period
  Interventions: Other: Normal Saline

INTERVENTIONS:
Device: Silver Diamine Fluoride — Silver Diamine Fluoride (Advantage Arrest) for the experimental group
  Other Names: Advantage Arrest
  Arms: Silver Diamine Fluordie Application
Other: Normal Saline — Normal Saline for the control group
  Arms: Normal Saline

SUMMARY:
Gingivitis in the geriatric population is one of the growing global public health concerns, thus finding the most effective and non-invasive approach to prevent and treat gingivitis in the geriatric population is essential to prevent tooth loss and maintain oral health and function. Silver Diamine Fluoride (SDF) is Class II medical device. It was cleared for use in US August 2014 and became commercially available in April 2015. It is a chemical agent which has bifunctional properties. The silver itself kills caries causing bacteria directly. Silver and fluoride together interact to form fluorapatite, in addition, assist in hardening the teeth and preventing further demineralization.

Even though SDF has been approved in dental caries prevention and treatment, there are no published studies or evidence that evaluated the direct effect of SDF on gingivitis. If SDF improves or prevents gingivitis is unknown. The main goal of this clinical study is to investigate the effect of SDF on gingival status in geriatric patients with gingivitis. There is an urgent need to solve this common oral disease in the geriatric population. The logic for this research in a geriatric population is to find the most effective approach to treat gingivitis to prevent tooth loss and maintain oral health and function.

To find an effective approach to treat gingivitis in the geriatric group, we will investigate the effectiveness of SDF application on gingival tissues in this group. The patients with gingivitis will be randomly allocated to two groups: group1(case group) will receive SDF application and group 2 (control group) will receive a normal saline application. The gingiva will be evaluated for both groups at baseline before the application. Then 2 weeks and 4 weeks after the last application of the intervention. In addition, a sample of plaque will be taken from the teeth selected in this study by swab using the dental kit (Ubiome) before and after both applications to quantify the presence of bacterial pathogen at baseline and follow up visits. The feasibility of this proposed therapy is supported by published literature that has shown that SDF was effective in dental and root caries prevention and treatment in geriatric patients.

DETAILED DESCRIPTION:
The Aims

* Aim 1 To investigate the effect of SDF application on gingival status in elder patients with gingivitis. To accomplish this aim, the subjects with gingivitis will be randomly allocated to two groups: group 1(case group) will receive SDF application and group 2 (control group) will receive Normal Saline. The SDF and normal saline will apply on the selected teeth with gingivitis once a week during a three-week period. The gingival status will be evaluated at baseline before the application of either SDF or normal saline. Then at the second week and fourth week after the final application. The measurable outcomes will be Plaque Index (PI) and the Gingival Index (GI). In addition, record of existing brushing and flossing habits. If SDF application shows an improvement in the gingival condition (reduction in the plaque and gingival indices) in treatment group comparing to the control group it indicates that its effectiveness not only on dental caries as published, but it is also may extended to include gingivitis.
* Aim 2 To quantify the presence of bacterial pathogen in the dental biofilm. To accomplish this aim, a sample of dental plaque will be taken from the teeth selected in this study by swab using the dental kit (Ubiome) before and after the SDF or normal saline application to quantify the presence of bacterial pathogen at baseline before the application, 2 weeks and 4 weeks after the application.

Summary:

The proposed therapeutic intervention of Silver Diamine Fluoride (SDF) in treating geriatric patients with gingivitis will establish a new adjunctive and inexpensive protocol for treatment of gingivitis. Gingivitis is inflammation of gingival tissues caused by dental biofilm bacterial infection. Left untreated, gingivitis will cause tooth loss. The preliminary results will provide new recommendations for treating geriatric patients in a safe, effective, and low-cost manner. This study will also address the gap in scientific knowledge regarding the use of SDF to treat gingivitis in elderly patients.

Research Hypothesis: The application of SDF varnish is expected to improve the gingival condition and can be an effective approach in the treatment of gingivitis in geriatric patients.

Null Hypothesis: The application of SDF varnish does not improve the gingival condition and cannot be an effective approach in the treatment of gingivitis in geriatric patients.

Research Question: Does the application of silver Diamine Fluoride on teeth with gingivitis will improve the gingival condition in geriatric patients with gingivitis

ELIGIBILITY:
Inclusion Criteria:

* Age group 65 years and older
* Males and females
* Minimum of 6 remaining teeth with gingivitis (at least one posterior tooth should be present)
* Every participant should agree to not brush or floss three days prior the data collection
* Every participant should agree to not use any mouthwash or Fluoride treatment for the entire study period
* All socioeconomic status included

Exclusion Criteria:

* Active chemotherapy or radiotherapy
* Known history of allergy to Silver Particles
* Uncontrolled diabetes
* Use of antibiotics in the last three months
* Periodontal therapy in the last 3 months
* Mouth rinse such as Chlorhexidine (CHX) at least 30 days prior to the study
* Smoking
* Epileptic patients on medication cause gingival overgrowth
* Patients who are unable to give consent
* Teeth with periodontitis

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
The change in Gingival Index GI (for Gingival Inflammation) | Assessment of the change from the baseline at 2 weeks and 4 weeks after the final application of either Silver Diamine Fluoride or Chlorhexidine
  The change in Gingival Index GI (for Gingival Inflammation) from Baseline before the application of either Silver Diamine Fluoride or Chlorhexidine and at two weeks and four weeks after the final application of either Silver Diamine Fluoride or Chlorhexidine
The change in Plaque Index PI (for dental plaque accumulation) | Assessment of the change from the baseline at 2 weeks and 4 weeks after the final application of either Silver Diamine Fluoride or Chlorhexidine
  The change in Plaque Index PI (for dental plaque accumulation) from baseline before the application of either Silver Diamine Fluoride or Chlorhexidine and at two weeks and four weeks after the final application of either Silver Diamine Fluoride or Chlorhexidine

SECONDARY OUTCOMES:
Assessment of microbial counts in Dental Plaque | Three times evaluation at baseline before the application of the intervention, then at 2 weeks and 4 weeks after the final application of either Silver Diamine Fluoride or Chlorhexidine
  Dental Plaque sample taken from each participant, labeled and send to the lab for analysis of bacterial counts (using Ubiome dental kit)

CONTACTS AND LOCATIONS:
Overall Officials: WEDAD ALSHEHRI, BSDH, MS., Study Director — Texas A&M University College of Dentistry
Locations (2):
- United States (2):
  - Notre Dame Court (Seniors Independent Living), Dallas, Texas
  - Dickinson Place (Seniors Independent Living), Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noureldin A, Alshehri W, Tapias H, Mallonee L, Mancl LM, Milgrom P, Svboda K. Efficacy of 38% silver diamine fluoride in reducing gingival inflammation and plaque accumulation in older adults living in retirement-homes: A randomized controlled pilot trial. J Dent. 2024 Apr;143:104890. doi: 10.1016/j.jdent.2024.104890. Epub 2024 Feb 20. PMID 38387597